CLINICAL TRIAL: NCT02668172
Title: Efficacy and Safety of Pasireotide Long Acting Release (LAR) in Combination With Weekly Pegvisomant in Previously Controlled Acromegaly Patients on Combination Treatment of Long-Acting Somatostatin Analogues and Weekly Pegvisomant
Brief Title: Pasireotide LAR and Pegvisomant Study in Acromegaly
Acronym: PAPE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, s neggers, Consultant endocrinology, Erasmus Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL49517.078.14; 2014-002219-41 (EudraCT Number); NTR5282 (Registry Identifier: Dutch Trial Register)
Record Dates: First submitted 2015-12-07; First posted 2016-01-29 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Acromegaly
Keywords: pegvisomant; pasireotide LAR; long acting somatostatin analogues
MeSH Terms: conditions — Acromegaly | interventions — pasireotide; pegvisomant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pasireotide LAR 60 mg monotherapy week 12 (Experimental): After enrollment, acromegaly patients on combination treatment will half their regular weekly dose of pegvisomant (PEGV) for 12 weeks (run-in period).
  When insuline-like growth factor 1 (IGF-I) remains within the age adjusted normal limits after 12 weeks, PEGV and the LA-SSA (Octreotide Long Acting Release (LAR) or Lanreotide Autogel) with Pegvisomant (PEGV) are discontinued and patients are switched to pasireotide LAR 60 mg for 12 weeks.
  Interventions: Drug: Pasireotide LAR 60 mg
- Pasireotide LAR 60 mg and Pegvisomant week 12 (Experimental): When IGF-I rises above the adjusted normal limits after 12 weeks (run-in period), these subjects will switch their LA-SSA to Pasireotide LAR 60 mg every 4 weeks and continue with the reduced PEGV dose of the run-in period, for the remaining 12 weeks.
  Interventions: Drug: Pasireotide LAR 60 mg; Drug: Pegvisomant
- Pasireotide LAR 60 mg and Pegvisomant week 24 (Experimental): Between week 12 and 24 dose adaptations of PEGV are not permitted unless IGF-I drops below the age adjusted normal limits, then the dose of PEGV will be decreased stepwise with 20 mg weekly until IGF-I is within the age adjusted normal limits.
  At week 24, efficacy will be assessed, as the number of patients with a normal IGF-I in the two different groups; the combination Pasireotide LAR 60 mg / PEG V dose and monotherapy Pasireotide LAR 60 mg.
  From week 24 patients will continue with Pasireotide LAR 60 mg monotherapy, or Pasireotide LAR will be combined with 50% of the original dose of PEGV, or with an increasing dose of PEGV every 8 weeks depending on the treatment arm.
  Interventions: Drug: Pasireotide LAR 60 mg; Drug: Pegvisomant

INTERVENTIONS:
Drug: Pasireotide LAR 60 mg — as mono-therapy or in combination with pegvisomant
  Other Names: Signifor, SOM230
Drug: Pegvisomant — only in combination with pasireotide LAR
  Other Names: Somavert
  Arms: Pasireotide LAR 60 mg and Pegvisomant week 12; Pasireotide LAR 60 mg and Pegvisomant week 24

SUMMARY:
The objective of this study is to assess the efficacy of Pasireotide Long Acting Release (LAR) alone and in combination with weekly Pegvisomant (PEGV) in acromegaIy patients previously controlled with combination treatment of long-acting Somatostatin analogs (LA-SSAs) and PEGV.

DETAILED DESCRIPTION:
Pasireotide Long Acting Release (Signifor ®), a novel long-acting multi-receptor ligand somatostatin analogue, has been shown to be more effective for the treatment of GH-secreting pituitary adenomas than currently used long-acting somatostatin analogues (LA-SSAs). The long-term efficacy of acromegaly patients using LA-SSAs in combination with PEGV was over 90% in terms of normalization of IGF-I. The combination of PEGV with pasireotide LAR has not been studied yet. Combining PEGV with pasireotide LAR could result in a lower dose and less injections of pegvisomant. This may ultimately lead to a more cost-effective treatment and improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent male or female aged ≥ 18 years
* documentation supporting the diagnosis of acromegaly based on elevated GH and/or IGF-I levels due to a pituitary tumor
* the patient is treated with lanreotide Autogel or octreotide LAR and PEGV (twice) weekly for at least 6 months and has a serum IGF-I level within 120 % of the age adjusted normal limits. These patients were previously not controlled by somatostatin analogs alone.
* female of no childbearing potential or male. No childbearing potential is defined as being postmenopausal for at least 1 year, or women with documented infertility (natural or acquired) or using two acceptable contraceptive measures, except for oral contraceptives.
* male subjects must agree that, if their partner is at risk of becoming pregnant, they will use a medically accepted, effective method of contraception (i.e. use a condom) for the duration of the study
* subjects must be willing and able to comply with study restrictions and to remain at the clinic for the required duration during the study period and willing to return to the clinic for the follow up evaluation as specified in the protocol.

Exclusion Criteria:

Patients will not be included in the study if he or she:

* has undergone pituitary surgery or radiotherapy within 6 months prior to study entry.
* it is anticipated that the patient will receive pituitary surgery or radiotherapy during the study.
* has a history of hypersensitivity to lanreotide, octreotide or pegvisomant or drugs with a similar chemical structure
* has been treated with any unlicensed drug within the last 30 days before study entry.
* has abnormal hepatic function at study entry (defined as AST, ALT, gGT, alkaline phosphatase, or total bilirubin above 3 ULN)
* is at risk of pregnancy or is lactating. Females of childbearing potential must provide a negative pregnancy test within 5 days before the start of the study and must be using contraception. Non-childbearing potential is defined as post-menopause for at least one year, surgical sterilization or hysterectomy at least three months before the start of the study.
* has a history of, or known current problems with alcohol or drug abuse.
* has a mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study, and/or evidence of an uncooperative attitude.
* has abnormal baseline findings, any other medical condition(s) or laboratory findings that, in the opinion of the investigator, might jeopardize the subject's safety or decrease the chance of obtaining satisfactory data needed to achieve the objective(s) of the study.
* renal insufficiency, clearance < 50ml/min
* poorly controlled diabetes mellitus with an HbA1c > 9.0%
* patients with a QTc > 500 ms on the EKG
* participation in a clinical trial in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with normalized IGF1 levels at 24 weeks in the pasireotide LAR monotherapy group and in the pasireotide LAR combined with pegvisomant group | 24 weeks

SECONDARY OUTCOMES:
The proportion of patients with normalized IGF1 levels after 48 weeks of pasireotide LAR monotherapy | 48 weeks
The proportion of patients with normalized IGF1 levels after 48 weeks combination treatment of pasireotide LAR with weekly pegvisomant. | 48 weeks
The necessary dose of pegvisomant during combination treatment of pasireotide LAR with pegvisomant in patients with an IGF-I level within the age adjusted normal limits | 48 weeks
Change in tumor volume by pituitary MRI | Baseline and 48 weeks
Tolerability and safety profile of pasireotide Long Acting Release (LAR) monotherapy | 48 weeks
  Toxicity will be assessed using the National Cancer Institute-Common Toxicology Criteria Adverse Events version 4 (NCI-CTCAE v.4.03) and for laboratory assessments that include biochemistry, hematology, urinalysis; special safety assessments that include the regular monitoring and recording of blood glucose, insulin, HbA1c, GH and IGF-1, thyroid and liver function tests, gallbladder examinations and ECGs. Concomitant medications/Significant nondrug therapies will be assessed from study enrollment until the safety follow-up.
Tolerability and safety profile of pasireotide LAR and pegvisomant combination therapy | 48 weeks
  Toxicity will be assessed using the National Cancer Institute-Common Toxicology Criteria Adverse Events version 4 (NCI-CTCAE v.4.03) and for laboratory assessments that include biochemistry, hematology, urinalysis; special safety assessments that include the regular monitoring and recording of blood glucose, insulin, HbA1c, and IGF-1, thyroid and liver function tests, gallbladder examinations and ECGs. Concomitant medications/Significant nondrug therapies will be assessed from study enrollment until the safety follow-up.
Evaluation of long term effect of pasireotide LAR with or without pegvisomant on AcroQol, PASQ and signs and symptoms of acromegaly | Change in scores as measured by AcroQoL from baseline to week 48
  AcroQol is quality of life questionnaire specifically designed for acromegaly
Evaluation of long term effect of pasireotide LAR with or without pegvisomant on AcroQol, PASQ and signs and symptoms of acromegaly | Change in scores as measured by PASQ from baseline to week 48
  PASQ are questionnaire for the disease specific symptoms
Evaluation of long term effect of pasireotide LAR with or without pegvisomant on AcroQol, PASQ and signs and symptoms of acromegaly | Description of signs and symptoms of acromegaly
Evaluation of body composition by Dual-energy X-ray Absorptiometry (DEXA) scan | baseline and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Neggers, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Derived] Muhammad A, van der Lely AJ, Delhanty PJD, Dallenga AHG, Haitsma IK, Janssen JAMJL, Neggers SJCMM. Efficacy and Safety of Switching to Pasireotide in Patients With Acromegaly Controlled With Pegvisomant and First-Generation Somatostatin Analogues (PAPE Study). J Clin Endocrinol Metab. 2018 Feb 1;103(2):586-595. doi: 10.1210/jc.2017-02017. PMID 29155991
- See also: Summary of study at the WHO International Clinical Trials Registry Platform — http://apps.who.int/trialsearch/Trial2.aspx?TrialID=NTR5282